CLINICAL TRIAL: NCT01210300
Title: Exploring Taiwanese Womens' Decision-making Regarding Vaginal Birth After Caesarean Section
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Mei-Man Chen, Department of Nursing, Chang Gung Institute of Technology
Other Study IDs: 99038
Record Dates: First submitted 2010-09-26; First posted 2010-09-28 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Caesarean Section
Keywords: caesarean section; vaginal birth after caesarean section; repeat caesarean section; childbirth expectation; childbirth experience

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of caesarean section (CS) has increased globally. Taiwan's statistics report a higher incidence of repeat CS compared to vaginal birth after caesarean (VBAC). This is concerning, as repeat CS are associated with increased maternal morbidity and mortality, and neonatal respiratory problems. VBAC is an approach which reduces the likelihood of such birth complications. However, there is limited information about Taiwanese women's decision regarding VBAC and their participation in decision-making. There is also a gap in literature about information for women about CS and VBAC.

DETAILED DESCRIPTION:
Ajzen's Theory of Planned Behaviour will theoretically underpin the study. A qualitative descriptive design using purposive sampling of 20 Taiwanese pregnant women who have previously had a CS with a live baby will be recruited from Chang Gung Memorial Hospital in Taiwan. In-depth interviews will be carried out in three phases: (1) between 34 weeks to 38 weeks of women's pregnancy; (2) on the third day after childbirth; and (3) at the fourth week after birth, the end of confinement. Boyatzis' Data Driven approach will be adopted to thematically analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Have had a previous CS with a live baby
* Currently at 34 to 38 weeks of pregnancy
* Medically eligible for a VBAC
* Have chosen to have a natural birth
* 20 years old and over
* Able to converse in Mandarin and/or Taiwanese

Exclusion Criteria:

* Previous myomectomy
* Previous classical caesarean section
* Two previous caesarean section
* Pregnant with complications

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-06; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Man Chen, Principal Investigator — Department of Nursing, Chang Gung Institute of Technology
Locations (1):
- Chang Gung Institute of Technology, Taoyuan District, Taiwan